CLINICAL TRIAL: NCT06676124
Title: Modulation of MMP-9/NGAL Ratio in Diabetic Patients With Early Renal Dysfunction by Piper Crocatum Functional Foods
Brief Title: MMP-9/NGAL Modulation by Piper Crocatum in Early Diabetic Nephropathy
Acronym: MMP-9/NGAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Andina Setyawati, Assistant Professor of Medical Surgical Nursing, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROT-2024-UH; 1220/UN4.14.1/TP.01.02/2024 (Other Grant/Funding Number: Research and Community Service (LPPM) Universitas Hasanuddin)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Early Renal Dysfunction in Diabetes; Diabetic Nephropathy; Inflammation and Oxidative Stress in Diabetic Patients
Keywords: Early Renal Dysfunction; Diabetes Complications; Piper crocatum; Antioxidants; Anti-inflammatory; Renal Biomarkers; Functional Foods
MeSH Terms: conditions — Diabetic Nephropathies; Inflammation; Renal Insufficiency; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Two parallel groups: one group receives Piper crocatum cookies, and the other group receives placebo cookies for 12 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blinded. Participants, care providers, investigators, and outcomes assessors are all masked to group assignments. Cookies for both the intervention and placebo groups are identical in appearance, taste, and packaging to prevent any indication of group allocation. The randomization and coding were handled by an independent party, and group assignments were concealed using sealed, opaque envelopes. All study personnel involved in data collection, analysis, and monitoring were also blinded to maintain the integrity of the results and minimize bias throughout the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piper crocatum Cookie Group (Experimental): Participants in this group will receive bioactive-rich cookies containing Piper crocatum extract, known for its antioxidant and anti-inflammatory properties. They will consume two cookies daily for 12 weeks, each formulated with a standardized 10% concentration of the ethyl acetate fraction of Piper crocatum extract. The intervention aims to modulate renal biomarkers associated with diabetic nephropathy
  Interventions: Dietary Supplement: Piper crocatum Extract Cookie
- Placebo Cookie Group (Placebo Comparator): Participants in this group will receive placebo cookies that are identical in appearance, taste, and texture to the Piper crocatum cookies but do not contain the active Piper crocatum extract. They will consume two cookies daily for 12 weeks. This group serves as a comparison to evaluate the effects of the Piper crocatum extract in the intervention group
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Piper crocatum Extract Cookie — Participants in the intervention group will receive cookies containing a standardized 10% ethyl acetate extract of Piper crocatum, known for its antioxidant and anti-inflammatory properties. These cookies will be consumed twice daily for 12 weeks. The intervention aims to assess the effects of Piper crocatum on renal biomarkers, such as MMP-9 and NGAL, in diabetic patients with early renal dysfunction
  Arms: Piper crocatum Cookie Group
Dietary Supplement: Placebo Comparator — Participants in the placebo group will receive cookies that are identical in appearance, taste, and texture to the active Piper crocatum cookies but do not contain the Piper crocatum extract. These cookies will be consumed twice daily for 12 weeks, serving as a control to assess the effects of the active intervention on renal biomarkers associated with diabetic nephropathy.
  Arms: Placebo Cookie Group

SUMMARY:
The goal of this clinical trial is to determine whether functional foods made with Piper crocatum (red betel leaf) can reduce kidney damage markers in people with diabetes who have early kidney dysfunction. Researchers aim to find out if these foods can help decrease inflammation and oxidative stress, which are known to worsen kidney problems in diabetes.

Participants are divided into two groups: one group will consume cookies containing Piper crocatum extract, while the other group will consume similar cookies without the extract (placebo). They will eat these cookies twice a day for 12 weeks.

This study will measure changes in two main kidney damage markers-MMP-9 and NGAL-before and after the intervention to see if Piper crocatum helps lower these markers and supports kidney health.

DETAILED DESCRIPTION:
This clinical trial investigates the potential of Piper crocatum-based functional foods to modulate renal biomarkers in diabetic patients with early renal dysfunction. Diabetic nephropathy, a common and severe complication of diabetes, is largely driven by chronic inflammation and oxidative stress. These conditions exacerbate renal damage and increase the risk of end-stage renal disease (ESRD). Current therapeutic approaches often fail to address these underlying inflammatory and oxidative pathways adequately, creating a need for complementary or alternative interventions.

Study Design and Intervention This study is a double-blind, randomized, placebo-controlled trial conducted in Indonesia. A total of 387 diabetic participants with early signs of renal dysfunction were recruited, and participants were randomly assigned to one of two groups: an intervention group and a placebo group. The intervention group receives cookies containing standardized extracts of Piper crocatum, a plant known for its high antioxidant and anti-inflammatory content, particularly flavonoids and glycoside polyphenols. The placebo group receives cookies identical in taste and appearance but without the active Piper crocatum ingredients.

Participants in both groups are instructed to consume two cookies per day for 12 weeks. The active cookies are carefully formulated to maintain bioactive integrity during production, ensuring that the concentration of Piper crocatum's key compounds is consistent and effective. The formulation includes 10% of an ethyl acetate fraction of Piper crocatum extract, chosen for its high antioxidant activity.

Objectives and Hypotheses The primary objective of this trial is to assess whether the consumption of Piper crocatum cookies reduces levels of matrix metalloproteinase-9 (MMP-9) and neutrophil gelatinase-associated lipocalin (NGAL) in diabetic patients with early renal dysfunction. MMP-9, an enzyme involved in extracellular matrix (ECM) remodeling, is a known marker for renal inflammation and fibrosis in diabetic nephropathy. NGAL, a marker of tubular injury, provides an indicator of oxidative stress and renal health. The secondary objective is to examine whether the MMP-9/NGAL ratio improves with Piper crocatum intervention, indicating a potential protective effect on both glomerular and tubular health.

Mechanism of Action and Prior Evidence The therapeutic action of Piper crocatum is hypothesized to involve the modulation of oxidative stress and inflammation through several key pathways. Flavonoids and glycoside polyphenols in Piper crocatum have demonstrated strong antioxidative properties, capable of scavenging free radicals and stabilizing cellular structures. These compounds also appear to influence regulatory proteins, including p53, SOD1, and E-cadherin, which play roles in cellular repair, apoptosis, and oxidative defense.

Recent studies have shown that Piper crocatum extracts can downregulate MMP-9 expression, thus preventing excessive ECM degradation and promoting tissue stability. Additionally, by reducing NGAL levels, Piper crocatum may protect against tubular injury, potentially lowering the risk of nephropathy progression. The current study expands on these findings by exploring Piper crocatum's effects specifically within a diabetic population with early renal dysfunction.

Biomarker Analysis Biomarker measurements for MMP-9 and NGAL will be conducted at baseline (Day 0) and after the 12-week intervention (Day 84). Blood samples will be collected following an 8-hour fasting period, and serum levels of MMP-9 and NGAL will be quantified using validated ELISA kits. These biomarker measurements provide a direct assessment of the intervention's impact on key pathways of renal injury and repair.

Statistical Methods The analysis will use both paired and independent statistical tests to compare biomarker levels between and within groups. The primary analysis will involve comparing the mean change in MMP-9, NGAL, and the MMP-9/NGAL ratio between the intervention and placebo groups. Effect sizes will be calculated to determine the magnitude of change associated with the Piper crocatum intervention. All statistical analyses will use a significance threshold of p < 0.05.

Expected Outcomes and Clinical Implications The anticipated outcome is a significant reduction in MMP-9, NGAL, and the MMP-9/NGAL ratio in the intervention group compared to the placebo group, indicating a potential protective effect on renal health. If successful, this study could establish Piper crocatum-based functional foods as a novel adjunct therapy for diabetic nephropathy, offering a dietary approach to mitigate the progression of renal dysfunction in diabetic populations.

By providing insights into a natural, bioactive intervention, this study may open new avenues for integrating functional foods into diabetic care to improve outcomes and enhance quality of life for patients at risk of advanced renal complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 20 years.
* Diagnosed with Diabetes Mellitus (DM).
* Serum urea levels above 43 mg/dL or serum creatinine levels above 0.90 mg/dL.

Exclusion Criteria:

* Pregnant or breastfeeding individuals.
* Patients with other medical conditions that require intensive care.
* Patients currently undergoing therapy for hypoalbuminemia.
* Known allergies to any ingredients in the study cookies.
* Other chronic conditions that might interfere with the study protocol (e.g., severe cardiovascular disease).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Change in MMP-9 and NGAL Levels in Diabetic Patients with Early Renal Dysfunction | Baseline and 12 weeks
  This measure evaluates the change in serum levels of matrix metalloproteinase-9 (MMP-9) and neutrophil gelatinase-associated lipocalin (NGAL) in diabetic patients with early renal dysfunction after 12 weeks of intervention. MMP-9 is associated with renal inflammation and extracellular matrix remodeling, while NGAL is a marker of tubular injury and oxidative stress. Blood samples will be collected at baseline and at the end of the 12-week period, and serum levels of MMP-9 and NGAL will be quantified using validated ELISA kits. This assessment aims to determine the potential effects of the Piper crocatum intervention on renal health by observing significant changes in these biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Center in Makassar, Indonesia, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be routinely shared to protect participant privacy and confidentiality. However, data may be made available to qualified researchers upon request, subject to approval by the study's principal investigator and in compliance with relevant privacy regulations and institutional policies.

REFERENCES:
- [Background] Serra R, Grande R, Butrico L, Buffone G, Calio FG, Squillace A, Rizzo BA, Massara M, Spinelli F, Ferrarese AG, de Caridi G, Gallelli L, de Franciscis S. Effects of a new nutraceutical substance on clinical and molecular parameters in patients with chronic venous ulceration. Int Wound J. 2016 Feb;13(1):88-96. doi: 10.1111/iwj.12240. Epub 2014 Feb 25. PMID 24612734
- [Background] Rojas-Quintero J, Wang X, Tipper J, Burkett PR, Zuniga J, Ashtekar AR, Polverino F, Rout A, Yambayev I, Hernandez C, Jimenez L, Ramirez G, Harrod KS, Owen CA. Matrix metalloproteinase-9 deficiency protects mice from severe influenza A viral infection. JCI Insight. 2018 Dec 20;3(24):e99022. doi: 10.1172/jci.insight.99022. PMID 30568032
- [Background] Rodriguez-Sanchez E, Navarro-Garcia JA, Aceves-Ripoll J, Abarca-Zabalia J, Susmozas-Sanchez A, Bada-Bosch T, Hernandez E, Merida-Herrero E, Andres A, Praga M, Fernandez-Ruiz M, Aguado JM, Segura J, Ruilope LM, Ruiz-Hurtado G. Variations in Circulating Active MMP-9 Levels During Renal Replacement Therapy. Biomolecules. 2020 Mar 26;10(4):505. doi: 10.3390/biom10040505. PMID 32225016
- [Background] Latronico T, Petraglia T, Sileo C, Bilancia D, Rossano R, Liuzzi GM. Inhibition of MMP-2 and MMP-9 by Dietary Antioxidants in THP-1 Macrophages and Sera from Patients with Breast Cancer. Molecules. 2024 Apr 10;29(8):1718. doi: 10.3390/molecules29081718. PMID 38675538
- [Background] Kumar M, Dev S, Khalid MU, Siddenthi SM, Noman M, John C, Akubuiro C, Haider A, Rani R, Kashif M, Varrassi G, Khatri M, Kumar S, Mohamad T. The Bidirectional Link Between Diabetes and Kidney Disease: Mechanisms and Management. Cureus. 2023 Sep 20;15(9):e45615. doi: 10.7759/cureus.45615. eCollection 2023 Sep. PMID 37868469
- [Background] Jones JI, Nguyen TT, Peng Z, Chang M. Targeting MMP-9 in Diabetic Foot Ulcers. Pharmaceuticals (Basel). 2019 May 22;12(2):79. doi: 10.3390/ph12020079. PMID 31121851
- [Result] Setyawati A, Wahyuningsih MSH, Nugrahaningsih DAA, Effendy C, Fneish F, Fortwengel G. Piper crocatum Ruiz & Pav. ameliorates wound healing through p53, E-cadherin and SOD1 pathways on wounded hyperglycemia fibroblasts. Saudi J Biol Sci. 2021 Dec;28(12):7257-7268. doi: 10.1016/j.sjbs.2021.08.039. Epub 2021 Aug 19. PMID 34867030
- [Result] Setyawati A, Saleh A, Tahir T, Yusuf S, Syahrul S, Aminuddin A, Raihan M, Jafar N, Hamzah H, Arfian N. Matrix Metalloproteinase-9 Testing of Golden Rice Cookies With Piper Crocatum Active Extract for Preventing Foot Ulcers in Patients With Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 29;13:e49940. doi: 10.2196/49940. PMID 38422498
- [Result] Papadopoulou-Marketou N, Whiss PA, Eriksson AC, Hyllienmark L, Papassotiriou I, Wahlberg J. Plasma levels of tissue inhibitor of metalloproteinase-1 in patients with type 1 diabetes mellitus associate with early diabetic neuropathy and nephropathy. Diab Vasc Dis Res. 2021 Mar-Apr;18(2):14791641211002470. doi: 10.1177/14791641211002470. PMID 33775157
- [Result] Pan SC, Li CY, Kuo CY, Kuo YZ, Fang WY, Huang YH, Hsieh TC, Kao HY, Kuo Y, Kang YR, Tsai WC, Tsai ST, Wu LW. The p53-S100A2 Positive Feedback Loop Negatively Regulates Epithelialization in Cutaneous Wound Healing. Sci Rep. 2018 Apr 3;8(1):5458. doi: 10.1038/s41598-018-23697-5. PMID 29615682
- [Result] Nevo A, Armaly Z, Abd El Kadir A, Douvdevani A, Tovbin D. Elevated Neutrophil Gelatinase Lipocalin Levels Are Associated With Increased Oxidative Stress in Hemodialysis Patients. J Clin Med Res. 2018 Jun;10(6):461-465. doi: 10.14740/jocmr3360w. Epub 2018 Apr 13. PMID 29707087
- [Result] Danquah M, Owiredu WKBA, Jnr BAE, Serwaa D, Odame Anto E, Peprah MO, Obirikorang C, Fondjo LA. Diagnostic value of neutrophil gelatinase-associated lipocalin (NGAL) as an early biomarker for detection of renal failure in hypertensives: a case-control study in a regional hospital in Ghana. BMC Nephrol. 2023 Apr 26;24(1):114. doi: 10.1186/s12882-023-03120-6. PMID 37101162
- [Result] Bae MJ, Karadeniz F, Oh JH, Yu GH, Jang MS, Nam KH, Seo Y, Kong CS. MMP-Inhibitory Effects of Flavonoid Glycosides from Edible Medicinal Halophyte Limonium tetragonum. Evid Based Complement Alternat Med. 2017;2017:6750274. doi: 10.1155/2017/6750274. Epub 2017 Sep 20. PMID 29234420
- [Result] Alsawaf S, Alnuaimi F, Afzal S, Thomas RM, Chelakkot AL, Ramadan WS, Hodeify R, Matar R, Merheb M, Siddiqui SS, Vazhappilly CG. Plant Flavonoids on Oxidative Stress-Mediated Kidney Inflammation. Biology (Basel). 2022 Nov 26;11(12):1717. doi: 10.3390/biology11121717. PMID 36552226
- [Result] Kunadu AP, Aboagye EF, Colecraft EK, Otoo GE, Adjei MYB, Acquaah E, Afrifa-Anane E, Amissah JGN. Low Consumption of Indigenous Fresh Dairy Products in Ghana Attributed to Poor Hygienic Quality. J Food Prot. 2019 Feb;82(2):276-286. doi: 10.4315/0362-028X.JFP-18-146. PMID 30682266
- See also: This study examines the effect of Piper crocatum-enriched Golden Rice cookies on diabetic foot ulcer prevention by modulating MMP-9 levels. The cookies are designed to reduce inflammation and support diabetic foot health through dietary intervention — https://pubmed.ncbi.nlm.nih.gov/38422498/